CLINICAL TRIAL: NCT03139279
Title: Comparing Time to Readiness for Discharge After Colonoscopy: Propofol and Dexmedetomidine vs Propofol Only Sedation
Brief Title: Propofol and Dexmedetomidine Versus a Propofol Only Regimen for Sedation During Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York - Downstate Medical Center (Other)
Responsible Party: Principal Investigator, Dennis Dimaculangan, Clinical Associate Professor, State University of New York - Downstate Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB: 932304
Record Dates: First submitted 2017-04-24; First posted 2017-05-03 (Actual); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Colonoscopy
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine and propofol (Experimental): Intravenous dexmedetomidine 0.3 ug/kg followed by propofol. Titrated doses of propofol will be given at the discretion of the anesthesiologist based on a target BIS range between 60-70.
  Interventions: Drug: Dexmedetomidine; Drug: Propofol
- Saline placebo and propofol (Placebo Comparator): Intravenous saline placebo followed by propofol. Titrated doses of propofol will be given at the discretion of the anesthesiologist based on a target BIS range between 60-70.
  Interventions: Other: Saline placebo; Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 0.3 ug/kg intravenous bolus
  Other Names: Dex; Precedex
  Arms: Dexmedetomidine and propofol
Other: Saline placebo — Intravenous saline/placebo
  Arms: Saline placebo and propofol
Drug: Propofol — Propofol titrated intravenous boluses
  Other Names: Diprivan

SUMMARY:
An ideal sedative for colonoscopy should have properties that include: rapid onset and offset of action, provide cardiopulmonary stability, have minimal adverse effects, and allow for smooth recovery, and early discharge. Propofol is often used solely because of its rapid onset and short duration of action---a property which is ideal for a fast recovery and early discharge in the ambulatory setting. However, the use of propofol has been associated with undesirable effects such as hypotension, hypoventilation and apnea requiring assisted ventilation.

Balanced anesthesia, using a combination of medications with different mechanisms of action can reduce the total amount of each sedative agent used and minimize their side effects while achieving the desired level of sedation. Dexmedetomidine is one agent that has been used either alone or in combination with propofol for sedation during colonoscopy. While there are many advantages to using dexmedetomidine, there is concern that the use of this agent for sedation during colonoscopy may prolong post-operative recovery time and readiness for discharge home.

No study has definitively assessed whether the use of dexmedetomidine in combination with propofol during ambulatory colonoscopy prolongs post-operative recovery time as determined by the Modified Post Anesthesia Discharge Scoring System (MPADSS).

DETAILED DESCRIPTION:
In this study, investigators plan to prospectively compare in a randomized, controlled, double-blind trial, the sedation technique for colonoscopy between two groups. Group 1: sedation with dexmedetomidine and propopfol versus group 2: sedation with saline placebo and propofol.

The study will have the following outcome measures for each group.

Primary outcome measure:

Readiness-for-discharge (RFD) at 10, 20 and 30 minutes after the colonoscopic procedure. Ready-for-discharge is defined as attainment of MPADSS score of 9-10.

Secondary outcome measures:

1. Total propofol consumption in mg/kg/duration of procedure in minutes;
2. Side effects:

   1. lowest intraoperative percent (%) drop in mean arterial pressure (MAP) from baseline,
   2. incidence of sustained bradycardic episodes (HR<50 for at least 5 minutes) intraoperatively,
   3. incidence of apneic episodes intraoperatively requiring positive pressure ventilation.

Methods:

One hundred patients will be recruited and randomized into two groups. For sedation, Group 1 will receive intravenous dexmedetomidine 0.3 ug/kg bolused at the onset of the procedure followed by titrated doses of propofol. Group 2 will receive a saline placebo bolus at the onset of the procedure followed by titrated doses of propofol. A hospital research pharmacist, based on a randomization table, will allocate to the anesthesia provider giving the sedation, the bolus syringe labelled dexmedetomidine/or saline study agent. The anesthesia provider, gastroenterologist, nurses as well as the subject will be blinded as to the syringe's actual content. A Bispectral Index (BIS) Monitor will be used during sedation. All subjects will be targeted to maintain a BIS score between 60-70. Outcome measures will be evaluated for statistical significance in a non-inferiority assessment.

Investigators hypothesize that there will be no difference in the time to discharge between the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

• patients scheduled to undergo colonoscopy at SUNY Downstate Medical Center.

Exclusion Criteria:

* < 18 years old
* > 75 years old
* Cognitively Impaired patients (Cognitively impaired patients are excluded from the study because our primary outcome involves a very strict discharge criteria that requires the patient to respond to and perform tasks on our pre-existing discharge scale checklist. These may be impossible to assess or will be difficult to standardize for patients whom are Cognitively Impaired.)
* Pregnant patients
* Patients who use a wheelchair or ambulates with crutches (Patients using a wheelchair are excluded from the study because our primary outcome involves a very strict discharge criteria that requires the patient to respond to and perform tasks on our pre-existing discharge scale checklist. These may be impossible to assess or will be difficult to standardize for patients whom who use a wheel-chair).
* Limited exercise tolerance (as this could represent active coronary disease)
* Total body weight greater than 105 kg (due to maximal dose of drug available in randomized syringes containing study drug)
* Propofol, soy, glycerol or dexmedetomidine allergy
* Significant renal impairment
* Significant hepatic impairment
* Inability to read or write in English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Dimaculangan, MD, Principal Investigator — SUNY Downstate Medical Center Department of Anesthesiology
Locations (1):
- SUNY Downstate Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vicari JJ. Sedation and analgesia. Gastrointest Endosc Clin N Am. 2002 Apr;12(2):297-311, viii. doi: 10.1016/s1052-5157(01)00011-3. PMID 12180162
- [Background] Faigel DO, Baron TH, Goldstein JL, Hirota WK, Jacobson BC, Johanson JF, Leighton JA, Mallery JS, Peterson KA, Waring JP, Fanelli RD, Wheeler-Harbaugh J; Standards Practice Committe, American Society for Gastrointestinal Endoscopy. Guidelines for the use of deep sedation and anesthesia for GI endoscopy. Gastrointest Endosc. 2002 Nov;56(5):613-7. doi: 10.1016/s0016-5107(02)70104-1. No abstract available. PMID 12397263
- [Background] Waring JP, Baron TH, Hirota WK, Goldstein JL, Jacobson BC, Leighton JA, Mallery JS, Faigel DO; American Society for Gastrointestinal Endoscopy, Standards of Practice Committee. Guidelines for conscious sedation and monitoring during gastrointestinal endoscopy. Gastrointest Endosc. 2003 Sep;58(3):317-22. doi: 10.1067/s0016-5107(03)00001-4. PMID 14528201
- [Background] Akarsu Ayazoglu T, Polat E, Bolat C, Yasar NF, Duman U, Akbulut S, Yol S. Comparison of propofol-based sedation regimens administered during colonoscopy. Rev Med Chil. 2013 Apr;141(4):477-85. doi: 10.4067/S0034-98872013000400009. PMID 23900369
- [Background] Tuncali B, Pekcan YO, Celebi A, Zeyneloglu P. Addition of low-dose ketamine to midazolam-fentanyl-propofol-based sedation for colonoscopy: a randomized, double-blind, controlled trial. J Clin Anesth. 2015 Jun;27(4):301-6. doi: 10.1016/j.jclinane.2015.03.017. Epub 2015 Mar 20. PMID 25801162
- [Background] Kamibayashi T, Maze M. Clinical uses of alpha2 -adrenergic agonists. Anesthesiology. 2000 Nov;93(5):1345-9. doi: 10.1097/00000542-200011000-00030. No abstract available. PMID 11046225
- [Background] Taittonen MT, Kirvela OA, Aantaa R, Kanto JH. Effect of clonidine and dexmedetomidine premedication on perioperative oxygen consumption and haemodynamic state. Br J Anaesth. 1997 Apr;78(4):400-6. doi: 10.1093/bja/78.4.400. PMID 9135361
- [Background] Arain SR, Ebert TJ. The efficacy, side effects, and recovery characteristics of dexmedetomidine versus propofol when used for intraoperative sedation. Anesth Analg. 2002 Aug;95(2):461-6, table of contents. doi: 10.1097/00000539-200208000-00042. PMID 12145072
- [Background] Jalowiecki P, Rudner R, Gonciarz M, Kawecki P, Petelenz M, Dziurdzik P. Sole use of dexmedetomidine has limited utility for conscious sedation during outpatient colonoscopy. Anesthesiology. 2005 Aug;103(2):269-73. doi: 10.1097/00000542-200508000-00009. PMID 16052108
- [Background] Dere K, Sucullu I, Budak ET, Yeyen S, Filiz AI, Ozkan S, Dagli G. A comparison of dexmedetomidine versus midazolam for sedation, pain and hemodynamic control, during colonoscopy under conscious sedation. Eur J Anaesthesiol. 2010 Jul;27(7):648-52. doi: 10.1097/EJA.0b013e3283347bfe. PMID 20531094
- [Background] Palumbo P, Tellan G, Perotti B, Pacile MA, Vietri F, Illuminati G. Modified PADSS (Post Anaesthetic Discharge Scoring System) for monitoring outpatients discharge. Ann Ital Chir. 2013 Nov-Dec;84(6):661-5. PMID 23165318
- [Background] Aldrete JA, Kroulik D. A postanesthetic recovery score. Anesth Analg. 1970 Nov-Dec;49(6):924-34. No abstract available. PMID 5534693

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We consented 122 patients of which 8 were immediately excluded for the following reasons: procedure began prior to randomization (3), inclusion criteria not met (3), anesthesiologist declined (1), patient withdrew consent (1); 114 were randomized into the treatment and placebo groups.
Period: Overall Study
Arm/Group | Dexmedetomidine and Propofol | Saline Placebo and Propofol
Started | 58 | 56
Completed | 51 | 50
Not Completed | 7 | 6
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 5 | 4
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: 114 were randomized into the treatment and placebo groups. Seven additional patients in the propofol-dexmedetomidine group and 6 in the propofol-saline group were excluded. Final n = 101
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine and Propofol | Saline Placebo and Propofol | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Categorical [Count of Participants; unit: Participants] — Age measured in years
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 43 | 37 | 80
    >=65 years | 8 | 13 | 21
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [52 to 61] | 56 [48.8 to 65] | 56 [50 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 64
  Male | 20 | 17 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 45 | 42 | 87
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Weight [Median (Inter-Quartile Range); unit: kilograms] | 77 [66 to 88.2] | 83.5 [69.1 to 93.4] | 80 [69.85 to 92]
Height [Median (Inter-Quartile Range); unit: inches] | 65 [64 to 67] | 65 [64 to 68] | 65 [64 to 67]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 27.6 [23.7 to 30.9] | 28.5 [24.6 to 32.8] | 28.31 [24.58 to 31.62]
ASA Physical Status Classification System [Count of Participants; unit: Participants] — The American Society of Anesthesiologists (ASA) physical status (ASAPS) classification system was developed to offer clinicians a simple categorization of a patient's physiological status that can be helpful in predicting operative risk. Developed By: ASA House of Delegates/Executive Committee. Last Amended: October 15, 2014 (original approval: October 15, 2014). Includes 4 categories: ASA I, II, III, IV, V, VI. The addition of "E" to the ASAPS (e.g., ASA 2E) denotes an emergency surgical procedure.
  Participants
    ASA I: A normal healthy patient | 7 | 1 | 8
    ASA II: A patient with mild systemic disease | 33 | 32 | 65
    ASA III: A patient with severe systemic disease | 11 | 17 | 28
    ASA IV: systemic disease, constant threat to life | 0 | 0 | 0
    ASA V: moribund pt, will not survive w/o operation | 0 | 0 | 0
    ASA VI: declared brain-dead patient | 0 | 0 | 0
Systolic Blood Pressure [Median (Inter-Quartile Range); unit: mmHg] | 134 [125 to 144.5] | 140.5 [122.2 to 147.7] | 135 [124 to 146]
Diastolic Blood Pressure [Median (Inter-Quartile Range); unit: mmHg] | 82 [75 to 90.5] | 81 [73 to 90.75] | 81 [74 to 91]
Mean Arterial Pressure [Median (Inter-Quartile Range); unit: mmHg] | 99 [94 to 111] | 99 [91 to 111] | 99 [92 to 110.3]
Heart Rate [Median (Inter-Quartile Range); unit: beats per minute] | 72 [61.5 to 78] | 71 [62.5 to 81] | 71 [62 to 79]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Ready for Discharge in Each Group at 30 Minutes Post Procedure
Description: Each subject was assessed for readiness for discharge at 10, 20 and 30 minutes after the procedure, using the Modified Post-Anesthesia Discharge Scoring System (MPADSS). A subject getting an MPADS score of 9-10 is deemed ready for discharge. The percentage of subjects ready for discharge in each group at 10, 20 and 30 minutes will be measured as primary outcome.
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine and Propofol | Saline Placebo and Propofol
Number analyzed (Participants) | 51 | 50
Participants | 26 | 44

2. Secondary Outcome: Average Total Propofol Consumption Per Group
Description: Total propofol consumption per subject was measured as μg/kg/min of procedure in minutes. The average propofol consumption in each group will be measured as secondary outcome.
Time Frame: between 7 and 57 minutes (median 19 min)
Measure: Median (Inter-Quartile Range); unit: μg/kg/min
Arm/Group | Dexmedetomidine and Propofol | Saline Placebo and Propofol
Number analyzed (Participants) | 51 | 50
μg/kg/min | 140 [120 to 200] | 180 [130 to 240]

3. Secondary Outcome: Number of Participants With Sustained Bradycardic Episodes
Description: Incidence of sustained bradycardic episodes (HR<50 for at least 5 minutes) intraoperatively in each group
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine and Propofol | Saline Placebo and Propofol
Number analyzed (Participants) | 51 | 50
Participants
  Sustained bradycardia | 3 | 1
  No sustained bradycardia | 48 | 49

4. Secondary Outcome: Lowest Intraoperative % Change in MAP From Baseline
Description: Lowest intraoperative percent (%) change in mean arterial pressure (MAP) from baseline (average in each group)
Time Frame: 30 minutes
Measure: Mean (Inter-Quartile Range); unit: percentage change
Arm/Group | Dexmedetomidine and Propofol | Saline Placebo and Propofol
Number analyzed (Participants) | 51 | 50
percentage change | 30 [25 to 38] | 21 [14 to 29]

5. Secondary Outcome: Number of Participants With Apneic Episodes Intraoperatively Requiring Positive Pressure Ventilation
Description: Incidence of apneic episodes intraoperatively requiring positive pressure ventilation in each group
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine and Propofol | Saline Placebo and Propofol
Number analyzed (Participants) | 51 | 50
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From patient enrollment through discharge from PACU
Description: The definition of adverse event, used to collect adverse event information in the study, did not differ from the clinicaltrials.gov.
  Additional information: list of potential adverse events relevant to the study included:
  * episodes of sustained bradycardia (greater than 5 minutes) associated with hypotension (MAP < 60 mm Hg) that were unresponsive to treatment. We used a cutoff of < 50 bpm to define bradycardia in this study.
  * apnea requiring positive pressure ventilation
Arm/Group | Dexmedetomidine and Propofol | Saline Placebo and Propofol
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50
Other Adverse Events (participants affected / at risk) | 0/51 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT03139279/Prot_SAP_000.pdf